CLINICAL TRIAL: NCT07295587
Title: Assessment of the Impact of Headache on the Employee Population of Libbs Pharmaceutical Ltd.
Status: Enrolling by invitation | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB2405
Record Dates: First submitted 2025-12-04; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Migraine Headache; Migraine
Keywords: Migraine; headache; Dr.Cefaleia; Libbs
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Libbs´employees: All volunteer employees of Libbs Pharmaceuticals residing in all Brazilian regions will participate in this research. An online questionnaire will be applied to assess research subjects understanding of migraine and health habits.

SUMMARY:
The main objective of this study is to evaluate the impact of primary headaches using data previously collected in a healthcare program conducted by Libbs with its employees. The study aims to identify the main types of headaches, assess their impact on work and quality of life, describe treatment modalities and healthcare services used, and analyze possible correlations between job position or sector and the occurrence of headaches, as well as their impact on productivity.

This retrospective observational study analyzes secondary data collected from Libbs employees during a healthcare program designed to understand the impact of migraine on work productivity and daily activities. Data were obtained through validated questionnaires made available via an app. As this study involves the analysis of previously collected data, it does not provide direct benefits to participants. However, it contributes to a better understanding of migraine symptoms among Libbs employees, supports awareness of the risks of self-medication, and highlights the effects of headaches on daily routines and productivity.

No therapeutic intervention is proposed in this study. Decisions regarding diagnosis, interventions, and treatments were made exclusively by the Dr. Cefaleia app team at the time of data collection, without any interference related to the development of this research. The HIT-6 score and the four WPAI outcomes will be analyzed: absenteeism (lost work time), presenteeism (impairment while working), overall work productivity loss (absenteeism plus presenteeism), and impairment in activities outside of work.

This study provides an opportunity to expand the understanding of the relationship between working conditions, headaches, health, and productivity. The analysis may help identify epidemiological patterns and occupational or social risk factors associated with headaches, supporting future preventive strategies and workplace health initiatives aimed at improving quality of life and productivity.

DETAILED DESCRIPTION:
Migraine has a major impact on quality of life and work capacity . In Brazil, although there are many studies on the prevalence of primary headaches, studies on the impact of this condition on work activities are still scarce. Recently, a cross-sectional study evaluated a large Brazilian cohort, providing important data on the impact of headache on quality of life, work, and use of health resources . However, this study focuses on the general population, including both workers and non-workers. There are still few studies that evaluate the impact of headache on work activities, relating the occurrence and intensity of headache and its impact on productivity to different job positions and hierarchical levels of workers.

Thus, given the high prevalence of migraine, its cost in terms of medical care, absenteeism, and impairment of social, family, and especially work activities, a more detailed study of this pathology in a population with high productive potential, such as employees of a national pharmaceutical industry, is urgently needed.

Although the clinical manifestations of migraine are well known, the impact of this condition on daily activities, especially in the workplace, is still widely underestimated. In this context, seeking to understand how migraine interferes not only with physical well-being, but also with the emotional, social, and professional dimensions of its employees' lives, Libbs promoted a healthcare program to assess health conditions related to migraine.

The assistance program used the Dr. Cefaleia para Médicos (Dr. Headache for Doctors) app with the following questionnaires: ID Migraine, in its validated Brazilian Portuguese version, the Headache Impact Test (HIT-6), also validated in Brazilian Portuguese, and the Brazilian migraine/headache impact questionnaire Work Productivity and Activity Impairment (WPAI). As previously mentioned, the WPAI is a tool that assesses the impact of health conditions, such as migraine, on work productivity and daily activities. The questionnaire included four main parameters:

1. Lost work time (absenteeism): Measures the time the individual was unable to work due to migraine.
2. Work impairment (presenteeism): Assesses the reduction in productivity while the individual is present at work but unable to perform their duties normally due to headache.
3. Overall productivity loss: Combines the effects of absenteeism and presenteeism.
4. Impairment of activities outside of work: Measures the impact of migraine on daily activities that are not related to work.

The objective of this research project is to perform statistical analysis of data already collected, without the need for additional primary data collection. Therefore, it will be conducted at the Libbs Farmacêutica LTDA office or remotely, from home.

To ensure the efficient and secure execution of the research, the team will have a private and reserved workspace, a stable and high-speed internet connection to facilitate communication between the team and remote access to the necessary database or storage system. Communication within the team will be carried out through platforms such as [Zoom, Microsoft Teams, Google Meet] for weekly meetings and discussions on the progress of the research.

The team will have computers with appropriate configurations and programs, which will ensure the necessary performance for data processing and analysis. Data protection will be a priority throughout the process. All data transferred to the Libbs team will be anonymized, and unauthorized access will be prevented. To ensure data integrity, periodic backups will be performed on secure servers, and the entire analysis process will comply with the General Personal Data Protection Law, with an emphasis on anonymization and security of personal data.

For this study, sociodemographic data (age, gender, education, position, sector, branch), presence of headache (yes or no), diagnosis, types of treatment, and scores from validated questionnaires, such as workLost, workCompromised, productivityLost, activityCompromised, and impact, collected during the assistance program carried out by Libbs with its employees, will be analyzed.

The collection of primary data did not involve the collection of directly identifiable personal information, so there will be no data such as name, document number, or other contact information that could identify participants, other than the email address, which was optional. For data whose email or other information allows for the indirect identification of individuals, a data anonymization process will be adopted to ensure that the information processed cannot be associated with specific individuals.

The anonymization technique adopted will be the removal or alteration of identifiable data through the following measures:

* Replacement of direct identifiers: if the database generated by the Dr. Cefaleia application contains any direct identifiers, these variables will be removed or replaced by random codes. These codes will be generated automatically and will have no relation to the original data that would allow the individual to be re-identified.
* Data grouping: Where possible, information will be grouped so that the individuality of each participant is not revealed. For example, variables related to age groups or job categories, department, or branch may be converted into ranges to avoid direct association with a specific individual.
* Variable generalization: Some variables that could be used to indirectly identify a person (such as job title, sector, branch, or details of very specific contexts) will be generalized, using, for example, broad categories to preserve anonymity.

These measures will ensure that the data used in the study cannot be associated with specific individuals, either directly or indirectly, in accordance with the principles of the General Personal Data Protection Law and the ethical standards applicable to research involving human subjects.

Anonymization will be performed by the researcher in charge before any analysis or sharing of data with Libbs, so that any information that allows re-identification will be permanently removed or modified, ensuring that participants remain anonymous and protected throughout the research process.

ELIGIBILITY:
Inclusion Criteria:

* This analysis will include data from all employees who participated in this assistance program and made their data available in the Dr. Cefaleia app.

Exclusion Criteria:

* Data from participants whose questionnaires were not completed in full will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Libbs´employees
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of migraine on Libbs employees | 1 month
  Given the observational nature of this study, the sample size for the study will not be calculated based on statistical considerations. Probabilistic and non-random sampling will be considered with the available data. The primary database contains data collected from 1,342 employees, out of a total of 2,957 employees at the company at the time. This is an observational, retrospective, descriptive study based on an anonymized secondary database, originating from data collected in a welfare program carried out by Libbs with its employees, who will response time on the form for entering data such as: age, gender, education, role, department, affiliate, presence of headache (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Renan B Domingues, Principal Investigator
Locations (1):
- Libbs Farmacêutica LTDA., São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Because the data is anonymized.